CLINICAL TRIAL: NCT05077033
Title: Treatment of Skin Tumours With Intratumoral Interleukin 12 Gene Electrotransfer in the Head and Neck Region
Brief Title: Intratumoral phIL12 GET
Acronym: SmartGeneH&N
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERIDEK-0086/2020
Record Dates: First submitted 2021-09-24; First posted 2021-10-13 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intratumoral phIL12 gene electrotransfer (Experimental)
  Interventions: Drug: phIL12 GET

INTERVENTIONS:
Drug: phIL12 GET — intratumoral phIL12 gene electrotransfer

SUMMARY:
Electroporation provides non-viral gene delivery method for plasmid DNA. Its clinical application was already proven in preclinical and in clinical trial in treatment of melanoma skin metastases with plasmid coding IL-12, in USA. Intratumoral gene transfer of plasmid coding for IL-12 has proven safe end effective, having good local tumour control and some evidence indicates on abscopal effect. The EU directives recommend the use of plasmids without the gene for antibiotic resistance. For this purpose we constructed plasmid coding for IL-12 in accordance with the EU regulatory requirements.

In the proposed study we intend to study the safety and tolerability of the constructed plasmid, phIL12, in treatment of basal cell carcinomas in patients with operable tumors in head and neck region. The study is designed as exploratory, dose escalating with the aim to determine the dose of plasmid that produces IL-12 expression in the tumours with best biological activity, infiltration of the immune cells and no toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, previously untreated cutaneous basal cell carcinoma located in head and neck region.
* Solitary tumors, with largest diameter up to 3 cm, in the region where curative surgery is feasible.
* Age 18-years or older.
* Life expectancy > 3 months.
* Physical performance in accordance with the Karnofsky scale ≥ 70 or < 2 in accordance with World Health Organization (WHO) scale.
* The patient must be capable of understanding the treatment procedure and possible adverse events, which may arise during treatment.
* The patient must be capable of signing the informed consent to participate in the clinical study (voluntary and conscientious consent after education).
* Prior to inclusion in the trial, the patient must be presented at a multidisciplinary advisory team meeting.

Exclusion Criteria:

* Known malignancy elsewhere in/on the body.
* Lesions not suitable for treatment with GET (invasion into the bone, infiltration of large vessels).
* A life-threatening infection and/or severe heart failure and/or liver failure and/or other life-threatening systemic diseases.
* Significantly reduced lung function, which requires the determination of DLCO. Patients should not be treated if DLCO is abnormal.
* Treatment with immunosuppressive drugs, steroids and other drugs that would affect poor wound healing.
* Age under 18-years.
* Major disruptions in the coagulation system (who does not respond to the standard therapy - replacement of vitamin K or freshly frozen plasma).
* A chronic decline in the kidney function (creatinine > 150 µmol/L).
* Epilepsy.
* Pregnancy and breast-feeding.
* The patient's incapability of comprehending the purpose or course of the trial, or not agreeing to be included in the trial.
* Patients unwilling or unable to comply with the protocol requirements and scheduled visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of acute adverse events | Adverse events 2 days after the treatment.
  CTCAE v.5.0 criteria
Number of adverse events 7 days after the treatment | Adverse events 7 days after the treatment.
  CTCAE v.5.0 criteria
Number of late adverse events | Adverse events 30 days after the treatment.
  CTCAE v.5.0 criteria
Evaluating quality of life with questionnaire one week after the treatment | Changes from baseline 7 days after the treatment.
  EORTC QLQ-C30
Evaluating quality of life with questionnaire one month after the treatment | Changes from baseline 30 days after the treatment.
  EORTC QLQ-C30

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Changes from baseline at 2, 7 and 30 days after the treatment.
  Determination of serum levels of IL-12 cytokine.
Concentrations of IL-12 and IFN-y in tumor samples | Changes from baseline at 7 and 30 days after the treatment.
  Determination of tumor IL-12 and IFN-y levels in tumor biopsies.

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Institute of Oncology Ljubljana, Ljubljana
  - University Medical Centre Ljubljana, Department of Otorhinolaryngology and Cervicofacial Surgery, Ljubljana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Groselj A, Bosnjak M, Jesenko T, Cemazar M, Markelc B, Strojan P, Sersa G. Treatment of skin tumors with intratumoral interleukin 12 gene electrotransfer in the head and neck region: a first-in-human clinical trial protocol. Radiol Oncol. 2022 Aug 14;56(3):398-408. doi: 10.2478/raon-2022-0021. PMID 35535423
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35535423/